CLINICAL TRIAL: NCT01071551
Title: The Impact of the "Nutrition Enrichment and Healthy Living Model" ( NEHLM) on Diet Quality.
Brief Title: The Impact of the "Nutrition Enrichment and Healthy Living Model" ( NEHLM) on Diet Quality, Physical Activity and Dental Health Among Children From Socioeconomically Disadvantaged Families in Beer Sheva
Acronym: NEHLM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Natalya Bilenko, Ben-Gurion University of the Negev Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SOR471208CTIL
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2009-11

CONDITIONS: Childhood Obesity
Keywords: Children; Obesity; Lifestyle; LSES; Caries
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle and health promotion (Experimental): The "Nutrition Enrichment and Healthy Living Model" (NEHLM) is an Integrative model covering variety of lifestyle issues such as nutrition, dental care, and physical activity. The model will be applied to kindergartens and a sample of their parents. Children participating will be given 10 lessons in nutrition, 5 lessons in dental-care and 20 physical activity lessons. Parents for children in this group will be given 2 nutrition-education meetings and a meeting with a dental clinician.2 additional meetings will be held for parents and children together, one in nutrition and one in dental-care.
  Interventions: Behavioral: Life-style intervention
- Physical activity only (Active Comparator): Children allocated to this group will attend physical activity classes only.
  Interventions: Behavioral: Physical activity only

INTERVENTIONS:
Behavioral: Life-style intervention — The "Nutrition Enrichment and Healthy Living Model" (NEHLM) is an Integrative model covering variety of lifestyle issues such as nutrition, dental care, and physical activity. The model will be applied to kindergartens and a sample of their parents. Children participating will be given 10 lessons in nutrition, 5 lessons in dental-care and 20 physical activity lessons. Parents for children in this group will be given 2 nutrition-education meetings and a meeting with a dental clinician.2 additional meetings will be held for parents and children together, one in nutrition and one in dental-care.
  Arms: Lifestyle and health promotion
Behavioral: Physical activity only — Children allocated to this group will attend 20 physical activity classes.
  Arms: Physical activity only

SUMMARY:
Childhood socioeconomic status (SES) is related to poor physical health, obesity, elevated cardiovascular risk factors and iron deficiency anemia. We plan to offer a comprehensive framework allowing the "Nutrition Enrichment and Healthy Living Model" (NEHLM) among a low SES Kindergarten children. The model offered is designed to take into account the current economic status of the child's family. We shall conduct a randomized controlled trial to assess the efficacy of the intervention.

Our main objective:

To compare the influence of the intervention on changes in food consumption, physical activity and ,and caries rates in the children in kindergartens where it is applied versus the control kindergartens.

The research hypothesis:

Integrative Nutrition Enrichment and Healthy Living Model (NEHLM) will improve health behaviors among children and parents in comparison to control intervention (physical activity only).

ELIGIBILITY:
Inclusion Criteria:

* Kindergarten children aged 4-7 Children from kindergartens defined as Low- SES population (by local municipality)
* Children whose parents agree to participate in the research

Exclusion Criteria:

* Children who suffer from any chronic disease
* Children who suffer from developmental problems
* Children who participate in a weight reduction treatment or program
* Children or parents who have any psychiatric problem or diagnosis

Ages: 48 Months to 84 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 258 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Children's weight and Height | Baseline, post intervention and at 4 months post intervention termination

SECONDARY OUTCOMES:
Caries rate (DMFT score) | Baseline, post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Natalya Bilenko, MD, M.PH, Principal Investigator — Ben Gurion Universty of the Negev Israel
Locations (1):
- Kindergardens, Beersheba, Israel

REFERENCES:
- [Derived] Kaufman-Shriqui V, Werbeloff N, Faroy M, Meiri G, Shahar DR, Fraser D, Novack Y, Bilenko N, Vardi H, Elhadad N, Pietrzak RH, Harpaz-Rotem I. Posttraumatic stress disorder among preschoolers exposed to ongoing missile attacks in the Gaza war. Depress Anxiety. 2013 May;30(5):425-31. doi: 10.1002/da.22121. PMID 23620192